CLINICAL TRIAL: NCT02732990
Title: Peripheral Metabolic Function in Chronic Heart Failure Patients: Key to Lessen the Cardiac Load
Brief Title: Peripheral Metabolic Function in Chronic Heart Failure Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anders Rasmussen Rinnov (Other)
Responsible Party: Sponsor-Investigator, Anders Rasmussen Rinnov, CIM administrator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: VEK-H-3-2013-048
Record Dates: First submitted 2014-11-06; First posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Heart Failure
Keywords: Training; One-legged exercise; Peripheral blood flow; Cardiac function; Muscle metaboreflex
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Exercise training - Whole body exercise (Experimental): Control subjects will train 2-legged cycling (whole body exercise) for 6 weeks
  Interventions: Behavioral: Exercise training
- Exercise training - One-legged exercise (Experimental): Control subjects will train high intense one-legged exercise for 6 weeks
  Interventions: Behavioral: Exercise training
- Exercise training - 2-legged cycling CHF (Experimental): CHF patients will train 2-legged cycling (whole body exercise) for 6 weeks
  Interventions: Behavioral: Exercise training
- Exercise training - CHF (Experimental): CHF Patients will train high intense one-legged exercise for 6 weeks
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — All gruoups will undergo 6 weeks of training intervention either with a small musclemass (one-legged exercise) or whole body exercise (two-legged cycling)

SUMMARY:
Exercise intolerance is a major limiting symptom in patients with CHF. However the poor correlation between the hemodynamic parameters of left ventricular performance at rest and exercise performance has led to the concept that peripheral factors such as muscle perfusion and muscle metabolism play a role as determinants of exercise capacity.

DETAILED DESCRIPTION:
The pathophysiology behind the breathlessness and fatigue experienced by CHF patients during exercise remains unclear. Recent evidence suggests that the peripheral skeletal muscle, which becomes abnormal in heart failure, is the source of afferent signals which disrupt normal patterns of cardiorespiratory control. When CHF patients exercise, an inappropriately strong sympathetic response further limits exercise tolerance by evoking larger than normal increases in peripheral sympathetic activation at a faster rate than in healthy individuals. A consequence of this exacerbated sympathetic response may be the further sympathetic restraint of blood flow to the active skeletal muscles resulting in hypoperfusion of the muscle vascular bed and fatigue. Small muscle mass exercise training increases muscle oxidative capacity and improves aerobic work capacity in CHF patients. A range of studies is proposed here that will provide an integrative view of the mechanistic basis behind exercise intolerance in CHF and relate the intramuscular metabolic status to the autonomic control of hemodynamics during exercise. An understanding of the mechanistic basis of the improved exercise tolerance with training, independent of improved resting cardiac function, will yield important information regarding the integrated control of blood flow and metabolic demand in CHF and highlight the importance of maintaining the integrity of the peripheral musculature in CHF.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association (NYHA) Class II - III
* Ejection fraction <35%
* Heart failure as a result of previous myocardial infarction
* Optimal treatment (ACE-inhibitors, beta-blockers)
* Stable heart failure
* Patients with and without implantable cardioverter defibrillator (ICD)

Exclusion Criteria:

* Peripheral vascular disease with symptoms of atherosclerosis (intermittent claudication)
* Aneurysm in a. femoral
* Moderate to severe heart valve disease
* Moderate to severe Chronic Obstructive Pulmonary Disease (COPD) with FEV1 <60%
* Heart Failure Patients with Biventricular pacemaker (BVP)
* Serious heart rhythm disturbances (arrhythmias such as atrial fibrillation and frequent premature ventricular contractions)
* Myocardial infarction within the last month
* Unstable angina (angina pectoris)
* Renal failure (creatinine greater than 2.5 mg / dL)
* Severe systemic disease of the nervous system, pulmonary or other severe organ involvement
* BMI> 30
* Pregnancy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline sympathetic nerve activity after 6 weeks of training | 6 weeks
  Sympathetic nerve activity, measured in plasma and dialysat with reference to nor-adrenaline.

SECONDARY OUTCOMES:
The effect of exercise training on exercise capacity in regards to oxygen uptake | 6 weeks
  Exercise capacity in regards to oxygen uptake (VO2peak) will be evaluated before and after the training intervention
The effect of exercise training on exercise capacity in regards to maximal workload | 6 weeks
  Exercise capacity in regards to Workload during 2-legged cycling (Wattpeak) will be evaluated before and after the training intervention
The effect of exercise training on exercise capacity in regards to a 6 min walk test | 6 weeks
  Exercise capacity in regards to a 6 min walk test (meters) will be evaluated before and after the training intervention

CONTACTS AND LOCATIONS:
Overall Officials: Stefan P Mortensen, Dr. Med, Study Chair — IMM - Department of Cardiovascular and Renal Research
Locations (1):
- Centre of Inflammation and Metabolism (CIM), Centre for Physical Activity Research, Copenhagen, Denmark